CLINICAL TRIAL: NCT03065205
Title: Breathing Counts: Evaluating Adherence in the Presence of Asthma Navigation Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-1845
Record Dates: First submitted 2016-08-25; First posted 2017-02-27 (Actual); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Patients will have adherence monitoring devices placed on their asthma inhalers (both daily and rescue medication). Adherence information will be sent to their PCP, specialist and school nurse monthly. Additionally, the navigator will speak with families every 2 months to discuss adherence data and address barriers.
  Interventions: Device: Propeller Health device + asthma navigator

INTERVENTIONS:
Device: Propeller Health device + asthma navigator — The patients will be monitored using the propeller health device for 6 months. The patients will be contacted at 2 month intervals by an asthma health educator to discuss barriers to adherence to asthma medications

SUMMARY:
To determine if an asthma navigator is helpful in improving communication between care providers and improving patient adherence to asthma medications after an asthma exacerbation.

DETAILED DESCRIPTION:
This study will aim to use technology to evaluate the effectiveness of a patient navigator for childhood asthma. The Investigators will place adherence monitoring devices on patient inhalers, and track use of patient asthma medicines. The Investigators will also utilize an asthma navigator who will discuss adherence with families and help to address any barriers to adherence that families identify. Additionally, the navigator will communicate patient specific adherence information to the patient's primary care physician (PCP) and school nurse. The adherence monitor will monitor communications between these providers.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years old,
* Admission to Children's Hospital Colorado with an asthma exacerbation between Jan 1 2017 and Dec 31 2017.

Exclusion Criteria:

* Language other than English or Spanish (application for monitoring adherence is only available in these languages)
* Presence of other complex medical problems including:

  * Cystic Fibrosis,
  * Tracheostomy/ventilator dependence,
  * other severe chronic lung disease, and
  * significant developmental delays.
* Home schooled or not in school
* Following up with an allergy or pulmonary provider outside the CHCO system after hospital discharge.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Hoch, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 65
Completed | 53
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.08 (2.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 18
  More than one race | 0
  Unknown or Not Reported | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Adherence of Use of Patient Asthma Inhalers
Description: Adherence will be measured via adherence monitoring devices for 6 months per patient. Change in device measured adherence from week 1 to week 24. Measured as change in average number of puffs of controller medication taken/puffs individually prescribed, measured between weeks 1 and 24.
Time Frame: Week 1 to Week 24
Population: Participants who were in the study for the 6 month period and had analyzable study data for at least 16 weeks of monitored time.
Measure: Median (Inter-Quartile Range); unit: Change in puffs taken/prescribed per wk
Arm/Group | Single Arm
Number analyzed (Participants) | 42
Change in puffs taken/prescribed per wk | -0.36 [-0.62 to -0.23]

2. Secondary Outcome: Degree of Asthma Control
Description: Measured via questionnaire data using Asthma Control Test (ACT) or Childhood Asthma Control Test (cACT) every 2 months. Reported at 6 months. Scores range from 5-25 on the ACT and 0-27 on the cACT. Scores >19 on either test indicate good asthma control
Time Frame: 6 months
Population: Total number of participants who responded to the 6 month survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 34
score on a scale
  Mean ACT score: number analyzed (Participants) | 8
  Mean ACT score | 20.6 (5.4)
  Mean cACT score: number analyzed (Participants) | 26
  Mean cACT score | 23.81 (3.23)

3. Secondary Outcome: Barriers to Adherence of Patient Asthma Inhalers
Description: Measured via questionnaire data obtained every 2 months. Reported at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 34
Participants
  Forgot | 15
  Felt child was better | 3
  Thought child didn't need it | 2
  Afraid inhaler could lead to addiction | 1
  Afraid inhaler could damage child | 1
  Side effects of inhaler | 1
  Inhaler not helping child | 1
  Didn't understand doctor's instructions | 0
  Thought method of application was too complicated | 0
  Child not cooperating with administration | 4
  Inhaler empty | 4
  Other reasons | 16

4. Secondary Outcome: Effectiveness of Communication Between Providers
Description: measured via survey to providers at the end of the intervention
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Provider Survey: This is a survey of providers that cared for participants in the study. We had a very low response rate for the exit survey.
Arm/Group | Provider Survey
Number analyzed (Participants) | 4
Participants
  Communication increased due to study | 1
  Communicated with other providers once or twice | 4

ADVERSE EVENTS:
Time Frame: 1 year
Description: Study staff received notifications on patients admitted to the ED or hospital and reviewed them for any connection to the device.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03065205/Prot_SAP_000.pdf